CLINICAL TRIAL: NCT04584957
Title: Prophylactic Negative Pressure Wound Therapy in Gynecologic Oncology: a Prospective Controlled Randomized Trial. (GO-VAC)
Brief Title: Prophylactic Negative Pressure Wound Therapy (VAC) in Gynecologic Oncology (G.O.)
Acronym: GO-VAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G.O-VAC. ID. 3316
Record Dates: First submitted 2020-09-18; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Wound Infection; Gynecologic Cancer
Keywords: Gynecologic oncologic laparotomic surgery; Prophylactic negative pressure wound therapy; Surgical site infection; Wound dehiscence
MeSH Terms: conditions — Wound Infection; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: After gynecologic oncologic laparotomic surgery and standard abdominal wall closure patients are randomized to one of the two arms of the study: sperimental arm (ciNPWT- closed incisional negative pressure wound therapy) and control arm (standard dressing)
Who Masked: Investigator
Masking Description: The investigator check the random list only when the patients is enrolled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAC therapy (Active Comparator): Prophylactic ciNPWT therapy positioning YES. Patients enrolled for placement of the device over a closed incision immediately post-operatively.
  Interventions: Device: VAC therapy
- Standard Closure (No Intervention): Prophylactic ciNPWT therapy positioning NO. Patients enrolled for standard laparotomic closure without ciNPWT positioning

INTERVENTIONS:
Device: VAC therapy — Prophylactic ciNPWT therapy (Prevena® KCI) entails placement of the device over a closed incision immediately post-operatively. Prevena® KCI may be left in place with no additional intervention for up to 7 days.
  Arms: VAC therapy

SUMMARY:
A prospective controlled randomized study aimed to prospectively evaluate, the impact and effectiveness of clean incision prophylactic vacuum negative pressure therapy on wound healing (ciNPWT) in women at high risk of developing wound complications who undergo major gynecologic surgery.

Gynecologic Oncology patients appear to be more at risk of developing wound complications than the general surgery population, reaching infection rates of 36 vs. 24 % that become 40 and 60% for obese and morbidly obese patients, respectively. Data about the use of ciNPWT are few, controversial and are of poor quality. No randomized, controlled trials have yet been reported in support of the use of ciNPWT in the gynecologic population.

DETAILED DESCRIPTION:
Wound complications in patients undergoing surgery for malignancies have a negative impact on quality of life and, in addition, are associated with an increase of the duration of hospital stay, imparting a significant socio-economic burden.

Several approaches have been proposed to reduce the wound complications rate without success. Instead, a novel and promising method has been employed which utilizes prophylactic negative pressure wound therapy placed over clean and closed surgical incisions immediately after surgery (ciNPWT).

In a recent meta-analysis across studies including all types of wounds and surgeries, ciNPWT was observed to reduce by 29.4 % the incidence of SSI and the odds of SSI. In the same meta-analysis, while limiting attention to general abdominal surgery alone, the weighted average of the selected studies reported a reduction in wound complications of 10.43% (13.54% vs 23.97%) for the ciNPWT group compared with controls which was a significant benefit.

This study is a prospective multi-centre controlled randomized trial, where after gynecologic oncologic laparotomic surgery and standard abdominal wall closure (if inclusion criteria result satisfied), patient is randomized to one of the two arms of the study: ARM A (sperimental): ciNPWT ARM B ( control): standard dressing.

For women in arm A: prophylactic ciNPWT therapy entails placement of the device over a closed incision immediately post-operatively. The device may be left in place with no additional intervention for up to 7 days. The use of the device does not require specialty care services or continued hospitalization. For women in arm B: standard dressing should be changed every 2 days after sterile medication.

People will be visited after 7 day of VAC-therapy (first visit) , discharge time (second visit or coincidence with the first visit), after 15 days from surgery (third visit for agraphis removal), after 30 days from surgery (fourth visit).

Sample size determination. A review of previous literature suggests that the incidence of wound-SSI is about 35% in G.O. patients. We assume that the use of ciNPWT could be linked to an wound-SSI incidence of 15% Setting a two-sided α=0.05 and power = 80%, the sample size is N=164 subjects. A dropout rate of 20% is added, reaching a final sample size of N=196 subjects (98 subjects per arm).

The primary objective will be achieved calculating and comparing the proportions of wound-SSI in the two arms. The comparison will be performed with a Chi-squared test. The same test will be applied to the comparisons of final and intermediate wound healing rates. The comparison of the proportion of wound complications and the proportion of patients in need of antibiotics will be achieved with a Chi-squared test, as well. Comparison of the time of operating room required to apply the dressings, hospital stay and time to adjuvant therapies will be performed with a T-test (if data are normally distributed) or with the Wilcoxon test (if data are not normal). A p-value <0.05 will be considered statistically significant.

All patient data will be collected and managed using an electronic database anonymously.

ELIGIBILITY:
Inclusion Criteria:

All patients subjected to midline incision (xiphoid-pubic/sub-xiphoid/umbilical-pubic incision) with:

* Moderate/Severe (Aletti score ≥3) Modified surgical complexity score in:

  * Ovarian cancer: primary debulking surgery (PDS) or interval debulking surgery (IDS) (minimum total hysterectomy+bilateral salpingo-oophorectomy+lymphadenectomy in early ovarian cancer [EOC] should be done to include the patient in the trial) or secondary debulking surgery at recurrence (SCS).
  * Endometrial cancer FIGO stage IV or staging surgery for high risk endometrial cancer
  * Uterine Sarcomas FIGO stage IIB-IV
  * Previous history of pelvic or abdominal radiotherapy (even locally advanced cervical cancer [LACC] post neoadjuvant (NAD) therapies [NAD chemo-radiation or chemotherapy alone])
  * Persistent or recurrent Cervical cancer
* Obesity (>30 Kg/sqm) in all Aletti score surgery and in all FIGO stage malignancies
* Controlled diabetes mellitus in all Aletti score surgery and all FIGO stage malignancies
* Heavy smokers ≥ 20 cigarettes a day in all Aletti score surgery and all FIGO stage malignancies.

Exclusion Criteria:

* uncontrolled diabetes mellitus
* severe cardiac dysfunction
* pregnancy
* underweight (body mass index [BMI] < 18.5 kg/sqm)
* long-term steroid use
* subcutaneous (e.g. Jackson Pratt) drainage positioning
* post-operative prophylactic use of antibiotics beyond the intraoperative short therapy
* contaminated (class III) and dirty/infected (class IV) incision [10]
* allergy to silver

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-09-18 (Estimated); Study Completion 2021-09-18 (Estimated)

PRIMARY OUTCOMES:
Change of the rate of surgical site infections at 15 days | 15 days
  To investigate whether the application of an ciNPWT device (Prevena Incision Management System, KCI, Inc., San Antonio, TX, USA) change the rate of surgical site infections (SSI) within 15 postoperative days in gynecologic oncology patients undergoing surgery, from 35 % to 15 %.

SECONDARY OUTCOMES:
Wound complications at 30 days | 30 days
  Evaluate, compare and describe wound complications through the systematic performing of surgical wound swab at 7, 15, 30 days after surgery
Change of the rate of surgical site infections at 7 days | 7 days
  Evaluate and compare the wound healing rate at intermediate evaluation
Estimated operative time | 1 day
  Evaluate and compare the time required for use of the operating room
Estimated hospital stay | 3-30 days
  Evaluate and compare the duration of hospital stay
Antibiotic therapy estimate | 30 days
  Evaluate and compare the proportions of patients requiring antibiotics because of wound complications
Time to start adjuvant therapy | 30-50 days
  Evaluate and compare the time to eventual adjuvant therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Professor, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS,Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Wechter ME, Pearlman MD, Hartmann KE. Reclosure of the disrupted laparotomy wound: a systematic review. Obstet Gynecol. 2005 Aug;106(2):376-83. doi: 10.1097/01.AOG.0000171114.75338.06. PMID 16055590
- [Background] Nugent EK, Hoff JT, Gao F, Massad LS, Case A, Zighelboim I, Mutch DG, Thaker PH. Wound complications after gynecologic cancer surgery. Gynecol Oncol. 2011 May 1;121(2):347-52. doi: 10.1016/j.ygyno.2011.01.026. Epub 2011 Feb 15. PMID 21324517
- [Background] Kim SI, Lim MC, Song YJ, Seo SS, Kang S, Park SY. Application of a subcutaneous negative pressure drain without subcutaneous suture: impact on wound healing in gynecologic surgery. Eur J Obstet Gynecol Reprod Biol. 2014 Feb;173:94-100. doi: 10.1016/j.ejogrb.2013.12.006. Epub 2013 Dec 15. PMID 24388401
- [Background] Kim SI, Lim MC, Bae HS, Shin SR, Seo SS, Kang S, Park SY. Benefit of negative pressure drain within surgical wound after cytoreductive surgery for ovarian cancer. Int J Gynecol Cancer. 2015 Jan;25(1):145-51. doi: 10.1097/IGC.0000000000000315. PMID 25386858
- [Background] Scalise A, Calamita R, Tartaglione C, Pierangeli M, Bolletta E, Gioacchini M, Gesuita R, Di Benedetto G. Improving wound healing and preventing surgical site complications of closed surgical incisions: a possible role of Incisional Negative Pressure Wound Therapy. A systematic review of the literature. Int Wound J. 2016 Dec;13(6):1260-1281. doi: 10.1111/iwj.12492. Epub 2015 Oct 1. PMID 26424609
- [Background] Willy C, Agarwal A, Andersen CA, Santis G, Gabriel A, Grauhan O, Guerra OM, Lipsky BA, Malas MB, Mathiesen LL, Singh DP, Reddy VS. Closed incision negative pressure therapy: international multidisciplinary consensus recommendations. Int Wound J. 2017 Apr;14(2):385-398. doi: 10.1111/iwj.12612. Epub 2016 May 12. PMID 27170231
- [Background] Semsarzadeh NN, Tadisina KK, Maddox J, Chopra K, Singh DP. Closed Incision Negative-Pressure Therapy Is Associated with Decreased Surgical-Site Infections: A Meta-Analysis. Plast Reconstr Surg. 2015 Sep;136(3):592-602. doi: 10.1097/PRS.0000000000001519. PMID 26313829
- [Background] Blackham AU, Farrah JP, McCoy TP, Schmidt BS, Shen P. Prevention of surgical site infections in high-risk patients with laparotomy incisions using negative-pressure therapy. Am J Surg. 2013 Jun;205(6):647-54. doi: 10.1016/j.amjsurg.2012.06.007. Epub 2013 Jan 30. PMID 23375758
- [Background] Lynam S, Mark KS, Temkin SM. Primary Placement of Incisional Negative Pressure Wound Therapy at Time of Laparotomy for Gynecologic Malignancies. Int J Gynecol Cancer. 2016 Oct;26(8):1525-9. doi: 10.1097/IGC.0000000000000792. PMID 27488215
- [Background] Mahdi H, Gojayev A, Buechel M, Knight J, SanMarco J, Lockhart D, Michener C, Moslemi-Kebria M. Surgical site infection in women undergoing surgery for gynecologic cancer. Int J Gynecol Cancer. 2014 May;24(4):779-86. doi: 10.1097/IGC.0000000000000126. PMID 24681712